CLINICAL TRIAL: NCT00989755
Title: An Evaluation of the Fax to Quit Program and Wisconsin Tobacco Quitline Utilization by Southeastern Wisconsin Clinics
Brief Title: Center for Disease Control (CDC) Fax to Quit/Academic Detailing Grant
Acronym: F2Q/EAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: M-2008-1335
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Smoking
Keywords: Tobacco dependence treatment in primary health care setting; Fax to Quit; Fax to Quit plus Enhanced Academic Detailing; Fax referral; Quitline
MeSH Terms: conditions — Smoking

ARMS (2):
- Fax to Quit plus Enhanced Academic Detailing (F2Q + EAD) (Experimental): Clinics in this group receive Fax to Quit materials and in person training from a Regional Outreach Specialist (ROS). The ROS also provides on-going training/technical assistance and performance feedback.
  Interventions: Other: Fax to Quit (F2Q)
- Fax to Quit alone (Placebo Comparator): Clinics in this group receive Fax to Quit materials and can download materials from a website.
  Interventions: Other: Fax to Quit (F2Q)

INTERVENTIONS:
Other: Fax to Quit (F2Q) — Clinics in this group receive electronic and hard copies of all materials necessary for implementing Fax to Quit within their clinics.

SUMMARY:
The purpose of this study is to evaluate Fax to Quit (F2Q) - a strategy that links state quitlines to health care delivery systems. FQ capitalizes upon the healthcare visit as an opportunity for intervention, consistent with the finding that approximately 70% of smokers visit a primary care physician each year. Successful integration of quitlines into healthcare delivery will transform regular healthcare visits into easily implemented, cost-beneficial avenues via which smokers all across America will be routinely inducted into effective cessation intervention. F2Q will be evaluated as follows:

1. Does F2Q increase contacts and "quality contacts," between the quitline and patients who smoke and receive health care at a participating clinic? A "quality contact" is defined as a quitline referral that results in the individual enrolling in the quitline counseling services. This aim will be assessed by measuring the rates of quitline referrals in 49 clinics before and after F2Q has been implemented.
2. Are contact rates and enrollment rates of F2Q increased by "Enhanced Academic Detailing" at clinic sites (with enhanced academic detailing comprising ongoing training/technical assistance as well as performance feedback)?
3. What are the features of the Fax to Quit (F2Q) and Fax to Quit plus Enhanced Academic Detailing (F2Q + EAD) interventions that key clinic personnel found helpful and easy to implement, as well as features that were unhelpful and difficult? This information will be gathered in qualitative assessments that also will identify clinic strategies and organizational features that facilitated successful implementation.
4. What are the incremental costs of instating and sustaining F2Q and F2Q + EAD and how do these costs compare to other quitline promotional strategies (e.g., paid media, medication give-away programs)?

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Smoker seeking medical care from general practice (internal medicine) clinic (clinic enrolled in study)
* Smoker motivated to make a quit attempt

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of Fax to Quit referrals | One year following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD MPH MBA, Principal Investigator — University of Wisconsin--CTRI
Locations (1):
- Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Sheffer MA, Baker TB, Fraser DL, Adsit RT, McAfee TA, Fiore MC. Fax referrals, academic detailing, and tobacco quitline use: a randomized trial. Am J Prev Med. 2012 Jan;42(1):21-8. doi: 10.1016/j.amepre.2011.08.028. PMID 22176842